CLINICAL TRIAL: NCT06939231
Title: Supporting University Students' Transition Towards Sustainable and Healthy Dietary Behaviours: A Living Lab Approach.
Brief Title: Supporting University Students Transition Towards Sustainable and Healthy Dietary Behaviours: A Living Lab Approach.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University College Dublin (Other)
Collaborators: PLAN'EAT Consortium (https://planeat-project.eu/) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: LS-23-72-Gibney.; 101061023 (Other Grant/Funding Number: European Union Horizon Europe)
Record Dates: First submitted 2025-03-05; First posted 2025-04-22 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Dietary Behaviours; Sustainable Healthy Diet; Personalised Nutrition
Keywords: Sustainable diet; Personalised nutrition; Dietary behaviours; University; Students; Living Lab

STUDY DESIGN:
Intervention Model Description: Sequential
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Living Lab approach to improve sustainable and healthy dietary behaviours. (Experimental): Living Lab baseline data collection measures, invitation to Study 1 and Study 2 and events/ activities (optional), and LL endpoint data collection measures.
  Interventions: Behavioral: Living Lab approach to improve sustainable and healthy dietary behaviours

INTERVENTIONS:
Behavioral: Living Lab approach to improve sustainable and healthy dietary behaviours — Living Lab baseline data collection measures, plus invitations to Study 1 and Study 2 and events/ activities (optional), and LL endpoint data collection measures.

SUMMARY:
The aim of this study is to test the efficacy, feasibility, and acceptability of the UCD PLAN'EAT Living Lab in promoting sustainable and healthy dietary behaviours among university students. This study will compare within participant changes in diet-related pre-specified outcomes (detailed below) at Living Lab baseline and endpoint and examine differences across participant engagement levels (e.g., low engagement versus high engagement) in Living Lab studies and events/ activities.

DETAILED DESCRIPTION:
The University College Dublin (UCD) Living Lab (LL) is a series of small studies designed to develop, implement, and evaluate strategies and interventions to support university students' transition towards a sustainable and healthy diet. The LL will use a participant-centred process involving established LL methodology, with stakeholders and students actively feeding into the study design. The baseline and endpoint data collection measures of the UCD PLAN'EAT LL are described in detail below, followed by an outline of a series of planned studies. The final design and outcome(s) of each will evolve as the LL progresses.

Two groups will be recruited to the UCD PLAN'EAT LL: a) UCD student participants, and b) stakeholder participants, on or connected to UCD Belfield Campus. Student and Stakeholder involvement in the LL is detailed separately below.

1. Student participants

   The LL study will recruit up to n=500 healthy students (aged 18-30 years) attending UCD Belfield Campus, to join the UCD PLAN'EAT LL Citizen panel. Upon successful screening and completion of informed consent, participants will be invited to join the UCD PLAN'EAT LL Citizen Panel, and then complete an initial baseline data collection, as described below. Following completion of baseline data collection measures, participants within the UCD PLAN'EAT LL Citizen Panel will subsequently be invited to participate in a series of studies (Study 1 and Study 2 detailed below), which will each form a separate registration. Students will also be invited to attend sustainable and healthy diet-related events/ activities. Following baseline data collection, subsequent participation in the LL series of studies (Study 1 and Study 2) and events/ activities is optional for all participants recruited to the UCD PLAN'EAT LL Citizen Panel.

   PLAN'EAT LL Citizen Panel Data Collection: LL Baseline

   Following informed consent, all participants recruited to the UCD PLAN'EAT LL Citizen Panel will be asked to complete a demographic, health, and lifestyle questionnaire, a diet-related questionnaire, and dietary assessment. The diet-related questionnaire will examine dietary attitudes and behaviours, including barriers and enablers to fruit and vegetables, legumes, meat, and high fat, salt, and sugar (HFSS) food consumption, nutrition knowledge, sustainable food literacy, self-efficacy, self-regulation, food neophobia, stage of change, and the self-report behavioural automaticity index. The dietary assessment will include: up to 3 online 24-hour dietary recalls (aim: 2 non-consecutive weekdays and 1 weekend day) via the web-based dietary recall tool, Foodbook24. All data will be collected using a secure online data collection platform.

   PLAN'EAT LL Citizen Panel Data Collection: LL Endpoint

   At the end of the overall LL study or when participants are completing their course of study at UCD, all participating students recruited to the PLAN'EAT LL Citizen Panel (detailed above) will be asked to complete a diet-related questionnaire and dietary assessment. The diet-related questionnaire will examine self-efficacy and the self-report behavioural automaticity index. The dietary assessment will include: up to 3 online 24-hour dietary recalls (aim: 2 non-consecutive weekdays and 1 weekend day) via the web-based dietary recall tool, Foodbook24. All data will be collected using a secure online data collection platform.

   UCD PLAN'EAT LL Citizen Panel Process Evaluation:

   At the end of the overarching LL study, UCD student participants will be invited to complete a study evaluation questionnaire. In addition, a subsample of UCD student participants will also be invited to participate in focus groups or one-to-one interviews at the end of the LL study. The evaluation questionnaire and focus groups/ interviews will explore topics encompassing, for example, their study experience, study acceptability, factors affecting participation rates (e.g., barriers and enablers), study engagement, perceived study effectiveness (e.g., evaluation on whether participants felt taking part in the Living Lab helped them to overcome the main barriers identified by the Living Lab student cohort to increasing fruit and vegetable intake, increasing legume intake, and reducing meat, and high fat, salt, and sugar (HFSS) food intake throughout the Living Lab study), and suggestions for improvement. The questionnaire and interviews will be guided by the Acceptability, Practicality, Effectiveness, Affordability, Spill-over effects, and Equity (APEASE) criteria. However, in line with the LL methodology, the evaluation details will be more fully articulated and confirmed as the LL study progresses.

   PLAN'EAT LL Citizen Panel Study 1: Behaviour-focused personalised nutrition intervention to promote sustainable and healthy diets in university students: a feasibility pilot study.

   The aim of Study 1 is to test the efficacy, feasibility, and acceptability of a novel, behaviour-focused personalised nutrition intervention compared to a control personalised nutrition intervention for improving adherence to sustainable and healthy diets in university students. This study has formed a separate registration (ClinicalTrials.gov ID: NCT06631469).

   PLAN'EAT LL Citizen Panel Study 2: A personalised nutrition intervention with tailored behavioural support to promote sustainable and healthy diets in university students.

   The aim of Study 2 is to test the efficacy of a novel personalised nutrition intervention with tailored behavioural support compared to a control personalised nutrition intervention (without tailored behavioural support) for improving adherence to sustainable and healthy diets in university students. Study 2 will incorporate key insights and learnings from Study 1 (including the process evaluation from Study 1). This study will form a separate registration.
2. Stakeholder participants

This UCD PLAN'EAT LL study will recruit n=20 stakeholders. Upon successful completion of informed consent, stakeholders will be regularly informally consulted at several time points throughout the duration of the LL study regarding their feedback and input on LL studies.

Process Evaluation:

At the end of the overarching LL study, stakeholders will be invited to participate in one-to-one semi-structured interviews to explore topics encompassing, for example, their study experience, study acceptability, factors affecting participation rates (e.g., barriers and enablers), study engagement, perceived study effectiveness, and suggestions for improvement. However, in line with the LL methodology, the evaluation details will be more fully articulated and confirmed as the LL study progresses. The interviews will be guided by the Acceptability, Practicality, Effectiveness, Affordability, Spill-over effects, and Equity (APEASE) criteria.

ELIGIBILITY:
Student participants:

Inclusion Criteria:

* Be a UCD student (aged 18-30 years) attending Belfield Campus.
* Be a healthy adult between the age of 18-30 years old, and in good general health.

Exclusion Criteria:

* Do not attend UCD Belfield Campus.
* Are under 18 years of age or over 30 years of age.
* Have a diagnosis of an acute or chronic medical condition that could interfere with the outcomes of the study. Such diagnoses include (but are not limited to) cardiovascular disease, diabetes mellitus, cancers (within the last 5 years), etc.

Stakeholder participants:

Inclusion Criteria:

- Stakeholder on or connected to UCD Campus.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 520 (Estimated)
Dates: Start 2024-02-26 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Living Lab: Legume intake (grams per day) | 32 months
  Student participants will record their diet at LL baseline (habitual diet) and LL endpoint (intervention diet) using an online 24-hour recall method. Legume intake will be calculated using dietary intake records (baseline: up to 3x 24-hour recalls; endpoint: up to 3x 24-hour recalls). The primary outcome measure is the change in legume intake (g/ day) as a result of the intervention.

SECONDARY OUTCOMES:
Living Lab: Plant-based food intake (grams per day) | 32 months
  Student participants will record their diet at LL baseline (habitual diet) and LL endpoint (intervention diet) using an online 24-hour recall method. Plant-based food intake will be calculated using dietary intake records (baseline: up to 3x 24-hour recalls; endpoint: up to 3x 24-hour recalls). The secondary outcome measure is the change in plant-based food intake (g/ day) as a result of the intervention.
Living Lab: Fruit intake (grams per day) | 32 months
  Student participants will record their diet at LL baseline (habitual diet) and LL endpoint (intervention diet) using an online 24-hour recall method. Fruit intake will be calculated using dietary intake records (baseline: up to 3x 24-hour recalls; endpoint: up to 3x 24-hour recalls). The secondary outcome measure is the change in fruit intake (g/ day) as a result of the intervention.
Living Lab: Vegetable intake (grams per day) | 32 months
  Student participants will record their diet at LL baseline (habitual diet) and LL endpoint (intervention diet) using an online 24-hour recall method. Vegetable intake will be calculated using dietary intake records (baseline: up to 3x 24-hour recalls; endpoint: up to 3x 24-hour recalls). The secondary outcome measure is the change in vegetable intake (g/ day) as a result of the intervention.
Living Lab: Meat intake (grams per day) | 32 months
  Student participants will record their diet at LL baseline (habitual diet) and LL endpoint (intervention diet) using an online 24-hour recall method. Meat intake will be calculated using dietary intake records (baseline: up to 3x 24-hour recalls; endpoint: up to 3x 24-hour recalls). The secondary outcome measure is the change in meat intake (g/ day) as a result of the intervention.
Living Lab: High fat, sugar, salt (HFSS) food intake (grams per day) | 32 months
  Student participants will record their diet at LL baseline (habitual diet) and LL endpoint (intervention diet) using an online 24-hour recall method. High fat, sugar, and salt food intake will be calculated using dietary intake records (baseline: up to 3x 24-hour recalls; endpoint: up to 3x 24-hour recalls). The secondary outcome measure is the change in high fat, sugar, and salt food intake (g/ day) as a result of the intervention.

OTHER OUTCOMES:
Living Lab: Diet-related greenhouse gas emissions reported as kilograms of carbon dioxide equivalents per day | 32 months
  Student participants will record their diet at LL baseline (habitual diet) and LL endpoint (intervention diet) using an online 24-hour recall method. Diet-related greenhouse gas emissions will be estimated using food, nutrient, and food-related greenhouse gas emission databases (measured as kilograms of carbon dioxide equivalents). The tertiary outcome measure is the change in diet-related greenhouse gas emissions (kgCO2-eq/day) as a result of the intervention.
Living Lab: Self-reported factors influencing sustainable and healthy dietary behaviours: Self-efficacy | 32 months
  Student participants will record their self-reported self-efficacy at LL baseline and LL endpoint via a questionnaire. Each participant's score can range from 8-40 (with 40 indicating greater self-efficacy). The quaternary outcome measure is the change in participants self-reported self-efficacy as a result of the intervention.
Living Lab: Self-reported factors influencing sustainable and healthy dietary behaviours: Self-reported behavioural automaticity index | 32 months
  Student participants will record their self-reported behavioural automaticity at LL baseline and LL endpoint via a questionnaire. Each participant's score can range from 4-28 (with 4 indicating low behavioural automaticity and 28 indicating high behavioural automaticity). The quaternary outcome measure is the change in participants self-reported behavioural automaticity as a result of the intervention.
Living Lab: Process Evaluation | 32 months
  At the end of the LL study, student participants will complete an evaluation questionnaire. Stakeholder participants and a subsample of student participants will be invited to participate in focus groups or one-to-one interviews. Participants will evaluate the Living Lab study on topics encompassing, for example, their study experience, study acceptability, factors affecting participation rates (e.g., barriers and enablers), study engagement, perceived study effectiveness, and suggestions for improvement. The questionnaire and focus groups/ interviews will be guided by the Acceptability, Practicality, Effectiveness, Affordability, Spill-over effects, and Equity (APEASE) criteria. The quinary outcome is stakeholder and student participants' evaluation of the LL study.
Living Lab Feasibility: Retention Rates | 32 months
  Following completion of Living Lab endpoint measures, retention rates (number of participants who complete endpoint measures / number of participants enrolled into the study x 100) will be calculated to assess study feasibility and acceptability.
Living Lab Feasibility: Data Completion Rates | 32 months
  Following completion of Living Lab endpoint measures, data completion rates (number of complete datasets for each outcome measure / number of participants enrolled × 100) will be calculated to assess study feasibility and acceptability.
Living Lab: Self-reported factors influencing sustainable and healthy diet consumption | 32 months
  Student participants will record their self-reported factors (barriers and enablers) influencing sustainable and healthy diet consumption to include the following food groups: fruit and vegetables, legumes, meat, and high fat, sugar, and salt (HFSS) foods, at LL baseline via a questionnaire. For each food group listed above, the questionnaire comprises twenty-two closed-response questions using a 5-point Likert scale (Score -2 (strongly disagree) to +2 (strongly agree)), and one open response question to ascertain any additional factors for each food group. Participants self-reported factors (barriers and enablers) influencing sustainable and healthy diet consumption for the following food groups: fruit and vegetables, legumes, meat, and HFSS foods will be analysed at baseline only to characterise university students' diet-related behaviours. Findings will inform future studies to be delivered within the Living Lab.
Living Lab: Self-reported factors influencing sustainable and healthy dietary behaviours: Self-regulation of eating behaviour | 32 months
  Student participants will record their self-reported self-regulation of eating behaviour at LL baseline via a questionnaire. Each participant's score can range from 5 to 25 (with 25 indicating greater self-regulation). Participants self-reported self-regulation will be analysed at baseline only to characterise university students' diet-related behaviours.
Living Lab: Self-reported factors influencing sustainable and healthy dietary behaviours: Food neophobia | 32 months
  Student participants will record their self-reported food neophobia at LL baseline via a questionnaire. Each participant's score can range from 10-70 (with 70 indicating greater food neophobia). Participants self-reported food neophobia will be analysed at baseline only to characterise university students' diet-related behaviours.
Living Lab: Self-reported factors influencing sustainable and healthy dietary behaviours: Nutritional knowledge | 32 months
  Student participants will record their self-reported nutritional knowledge at LL baseline via a questionnaire. Participant's nutritional knowledge scores will be calculated at LL baseline. A score of zero will be allocated for incorrect responses and a score of one will be allocated to each correct response and all scores will be summed (with higher scores indicating greater nutritional knowledge). Participants self-reported nutritional knowledge will be analysed at baseline only to characterise university students' diet-related behaviours.
Living Lab: Self-reported factors influencing sustainable and healthy dietary behaviours: Sustainable food literacy | 32 months
  Student participants will record their self-reported sustainable food literacy at LL baseline via a questionnaire. Participant's sustainable food literacy scores will be calculated at LL baseline. A score of zero will be allocated for incorrect responses and a score of one will be allocated to each correct response and all scores will be summed (with higher scores indicating greater sustainable food literacy). Participants self-reported sustainable food literacy will be analysed at baseline only to characterise university students' diet-related behaviours.

CONTACTS AND LOCATIONS:
Locations (1):
- University College Dublin, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: No
At the beginning of the study, each participant will have a study code assigned to them. All data collected from the study will be stored using these unique study codes. A file will be set up which will be stored in a separate location to the study data. This file will contain a list which will link each participants' contact details to the corresponding ID code. All stored information will be password-protected and only accessible to the research team/ named researchers on the project. At the end of the LL project, all data will be anonymised. Pseudonymised/ anonymised data will be shared with PLAN'EAT partners where appropriate.

REFERENCES:
- [Background] Appleton KM, McGill R, Neville C, Woodside JV. Barriers to increasing fruit and vegetable intakes in the older population of Northern Ireland: low levels of liking and low awareness of current recommendations. Public Health Nutr. 2010 Apr;13(4):514-21. doi: 10.1017/S1368980009991790. PMID 20230659
- [Background] Kliemann N, Wardle J, Johnson F, Croker H. Reliability and validity of a revised version of the General Nutrition Knowledge Questionnaire. Eur J Clin Nutr. 2016 Oct;70(10):1174-1180. doi: 10.1038/ejcn.2016.87. Epub 2016 Jun 1. PMID 27245211
- [Background] Gardner B, Abraham C, Lally P, de Bruijn GJ. Towards parsimony in habit measurement: testing the convergent and predictive validity of an automaticity subscale of the Self-Report Habit Index. Int J Behav Nutr Phys Act. 2012 Aug 30;9:102. doi: 10.1186/1479-5868-9-102. PMID 22935297
- [Background] Pliner P, Hobden K. Development of a scale to measure the trait of food neophobia in humans. Appetite. 1992 Oct;19(2):105-20. doi: 10.1016/0195-6663(92)90014-w. PMID 1489209
- [Background] Baungaard C, Lane KE, Richardson L. Understanding nutrition students' knowledge, perceived barriers and their views on the future role of nutritionists regarding sustainable diets. Nutr Bull. 2023 Dec;48(4):572-586. doi: 10.1111/nbu.12649. Epub 2023 Nov 10. PMID 37950523
- [Background] Kliemann N, Beeken RJ, Wardle J, Johnson F. Development and validation of the Self-Regulation of Eating Behaviour Questionnaire for adults. Int J Behav Nutr Phys Act. 2016 Aug 2;13:87. doi: 10.1186/s12966-016-0414-6. PMID 27484457
- [Background] Weller KE, Greene GW, Redding CA, Paiva AL, Lofgren I, Nash JT, Kobayashi H. Development and validation of green eating behaviors, stage of change, decisional balance, and self-efficacy scales in college students. J Nutr Educ Behav. 2014 Sep-Oct;46(5):324-33. doi: 10.1016/j.jneb.2014.01.002. Epub 2014 Mar 5. PMID 24613445